CLINICAL TRIAL: NCT05411406
Title: Proof-of-principle Study for the Prediction of Difficult Mask Ventilation Using 3D-Facescan and Machine Learning
Brief Title: Prediction of Difficult Mask Ventilation Using 3D-Facescan and Machine Learning
Acronym: MASCAN
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Institute of Medical Technology and Intelligent Systems at Hamburg University of Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-100811-BO-ff
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Mask Ventilation; General Anesthesia
Keywords: Risk prediction; Airway management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Patients undergoing ENT or OMS surgery with general anesthesia with facemask ventilation and tracheal intubation (observational)

SUMMARY:
The aim of this study is to prove feasibility and assess the diagnostic performance of a machine learning algorithm that relies on data from 3D-face scans with predefined motion-sequences and scenes (MASCAN algorithm), together with patient-specific meta-data for the prediction of difficult mask ventilation. A secondary aim of the study is to verify whether voice and breathing scans improve the performance of the algorithm. From the clinical point of view, we believe that an automated assessment would be beneficial, as it preserves time and health-care resources while acting observer-independent, thus providing a rational, reproducible risk estimation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduling for ENT or OMS surgery in general anaesthesia, who require facemask ventilation and tracheal intubation after induction of anesthesia
* Patients aged at least 18 years
* Ability to understand the patient information and to personally sign and date the informed consent to participate in the study
* The patient is co-operative and available for the entire study
* Provided informed consent/patient representative

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Rapid sequence induction or other contraindications for facemask ventilation
* Planned awake tracheal intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive sampling: Adult patients that undergo ENT or OMS surgery in a tertiary care hospital who require facemask ventilation and tracheal intubation after induction of anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Difficult facemask ventilation | 1 hour
  Observed difficult facemask ventilation after induction of anesthesia

SECONDARY OUTCOMES:
Difficult tracheal intubation | 1 hour
  Observed difficult intubation after induction of anesthesia
Difficult laryngoscopy | 1 hour
  Observed difficult laryngoscopy after induction of anesthesia
Number of attempts | 1 hour
  Observed during tracheal intubation
Failed direct laryngoscopy | 1 hour
  Observed during airwaymanagement
Cormack Lehane grade | 1 hour
  Grading of the best view obtained during laryngoscopy (I-IV)
Difficult mask ventilation alert | 1 hour
  Noted by the responsible anaesthesiologist after airway management
Difficult intubation alert | 1 hour
  Noted by the responsible anaesthesiologist after airway management
Intubation time | 1 hour
  Recorded during airwaymanagement
Time to sufficient mask ventilation | 1 hour
  Recorded during airwaymanagement
Classification of intubation difficulty | 1 hour
  VIDIAC score rating between -1 and 5 points
Percentage of glottis opening (POGO) | 1 hour
  Grading of the best view obtained during laryngoscopy (%)
Impossible facemask ventilation | 1 hour
  Observed impossible facemask ventilation after induction of anesthesia
Successful first attempt intubation | 1 hour
  Observed during airway management
Airway-related adverse events | 1 hour
  Laryngospasm, bronchospasm, larynx trauma, airway trauma, soft tissue trauma, oral bleeding, edema, dental damage, corticosteroid application, accidental esophageal intubation, aspiration, hypotension or hypoxia
Post-intubation recommendation for an intubation method | 1 hour
  Recommendation of the responsible anaesthesiologist after airwaymanagement
Minimal peripheral oxygen saturation (SpO2) | 1 hour
  Observed after induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany